CLINICAL TRIAL: NCT05074381
Title: Effect of Dry Needling of the M. Obliquus Capitis Inferior on Rotational Mobility and Headache Related Outcome Measures in Patients With Cervicogenic Headache: a Randomized, Controlled Experimental Study
Brief Title: Dry Needling of the M. Obliquus Capitis Inferior on Rotational Mobility and Headache Related Outcome Measures in CH.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-10474
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Neck Pain, Posterior; Headache; Mobility Limitation
Keywords: Dry Needling; Sham Needling; Myofascial Pain Syndrome; M. Obliquus Capitis Inferior
MeSH Terms: conditions — Neck Pain; Headache; Mobility Limitation; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): A single dry needling session will be performed with the subject lying in prone position. A trained physiotherapist will penetrate the needle into skin surface, fascia,into the muscle tissue at the MTrP location of the M. Obliquus Capitis Inferior, and will move the needle up and down to elicit local twitch responses.In case local twitch responses are elicited, this will be repeated until the local twitch responses are extinct. Afterwards, a rotational muscle energy technique will be applied to the atlanto-axial level.
  Interventions: Other: Dry Needling
- Sham needling (Sham Comparator): A single sham needling session will be performed with the subject lying in prone position. A trained physiotherapist will penetrate the needle into the skin surface at the MTrP location. The fascia and muscle tissue will not be penetrated. Afterwards, a rotational muscle energy technique will be applied to the atlanto-axial level.
  Interventions: Other: Sham Needling

INTERVENTIONS:
Other: Dry Needling — Dry needling (DN) is a myofascial treatment technique, in which a thin, solid filiform needle is inserted directly into the MTrP. During dry needling, local twitch responses (LTR) can be elicited. These are involuntary contractions of muscle fibers, leadi
  Arms: Dry needling
Other: Sham Needling — During sham needling, a solid, filiform needle is inserted in the skin surface at the trigger point location, without penetrating the fascia and muscle tissue.
  Arms: Sham needling

SUMMARY:
An experimental study will be conducted to evaluate the effect of dry needling on the M. Obliquus capitis inferior on rotational mobility and headache realted outcome measures in patients with cervicogenic headache.

DETAILED DESCRIPTION:
Headache is a common and disabling condition. Several primary and secondary headache forms have been described, such as migraine, tension-type headache and cervicogenic headache (CH). In patients with CH; we can see a reffered pain pattern to the head, possibly originating from a source in the (upper)cervical spine. It has been described that nociceptive input, originating from the C1-C3 nervous system may be responsible for pain referal to head and neck regions. Recently, the flexion-rotation test (FRT) has been described as one of the most usefel clinical tests in the clinical testing and research of CH. Other literature showed that the rotational movement during the FRT was diminished in patients with CH and these results were correlated to headache intensity. 5,6

To treat this disabling condition, manual therapy is already known to be an effective treatment strategy. However, the additional value of dry needling is still to be discussed. Since the M. Obliquus capitis inferior (M. OCI) finds its origin on the apex of the spinous processus of C2 and inserts on transverse processus of the atlas (C1); this muscle might be anatomically very relevant to influence rotational mobility in the upper cervical spine. Additionally, this muscle is responsible for proprioception and accurate positioning of the head and neck, due to the presence of a large amount of Golgi bodies and muscle spindles in the muscle. Considering the myofascial pain referal pattern of the M. OCI, a referred pain pattern to the temporal region may be present when active triggerpoints are present.

Previous research already showed some preliminary evidence for positive treatment effects by dry needling of the M. OCI in patients with cervicogenic dizziness and headache.

The goal of this study is to evaluate the effect of a single dry needling intervention of the M. OCI on rotational mobility and headache related parameters, in a group of cervicogenic headache patients with a positive flexion-rotation test (articular mobility test on level C1-C2).

In this experimental study, 40 patients with cervicogenic headache will be recruited. Participants are required to have complaints for at least 3 months. Participants are included based on online questionnaires, a clinical examination of neck and shoulder, and the identification of a MTrP in the M. OCI muscle. All participants will receive information and have to sign an informed consent form.

Participants will be subjected to baseline assessment, which involves questionnaires and measurements of the cervical spine.

Secondly, participants will be randomly allocated to either the dry needling group or a sham needling group. The dry needling group will receive a dry needling treatment at the identified trigger point location (M. OCI - heterolateral to the restricted rotationside) whereas the sham needling group will receive an intervention in which the needle only penetrates the skin but not the fascia and muscle tissue.

Rotational mobility will be evaluated after the needling intervention, afterwards all patients will receive a standardized manual therapy treatment (Muscle Energy Technique). Afterwards, all baseline measurements will be conducted again. This testing will be repeated one week after treatment as well.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervicogenic headache according to the ICHD-3 criteria:

A. Any headache fulfilling criterion C B. Clinical and/or imaging evidence1 of a disorder or lesion within the cervical spine or soft tissues of the neck, known to be able to cause headache2

C. Evidence of causation demonstrated by at least two of the following:

1. headache has developed in temporal relation to the onset of the cervical disorder or appearance of the lesion
2. headache has significantly improved or resolved in parallel with improvement in or resolution of the cervical disorder or lesion
3. cervical range of motion is reduced, and headache is made significantly worse by provocative manœuvres
4. headache is abolished following diagnostic blockade of a cervical structure or its nerve supply D. Not better accounted for by another ICHD-3 diagnosis3;4;5.

   * Age: 18-65 years
   * Headache for at least 1 day/week for at least 3 months
   * Limited mobility of the neck
   * Positive flexion-rotation test (<32 degrees on the left/right side or a difference of 10 degrees or more between left and right side)
   * NRS > 3/10

Exclusion Criteria:

* Primary headache forms: migraine, TTH
* Other secondary headaches that do not comply with the ICDH-3 criteria for CH
* Whiplash or other traumatic incident in the past
* Pregnancy or given birth in the last year
* Previous head, neck or shoulder surgery
* Cervical radiculopathy complaints
* Fear of needles
* Receiving other treatments for headache or neck pain (physical therapy/ostheopathy/chiropraxie...) in the previous month
* All possible contra-indications for dry needling (taking anti-coagulantia; infectional diseases; skin abnormalties in the head/neck-region; epilepsia; allergies for latex, nickel...)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Atlanto-axial rotational mobility after dry needling or sham needling assessed by the flexion-rotation test. | Baseline, Immediately after needling (DN or SN), immediately after manual therapy, 1 week after the needling intervention.
  Changes in Atlanto-axial rotational mobility after dry needling or sham needling will be assessed by the flexion-rotation test at baseline, immediately after needling (DN or SN); immediately after manual therapy and 1 week after treatment. Measurements will be registered with the digital EasyAngle Goniometer (Meloq).
  The change in Atlanto-axial rotational mobility after dry needling will be compared with the change Atlanto-axial rotational mobility after sham needling. Atlanto-axial rotational mobility be expressed in degrees.

SECONDARY OUTCOMES:
Changes in headache pain intensity | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Changes in pain score after dry needling, compared to sham needling, as assessed by the numeric rating scale (NRS).
  Subjects will have to report their actual pain complaints on a numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain) at baseline, immediately after dry or sham needling + manual therapy and 1 week after the intervention.
Changes in neck related disability | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Changes in neck disability scores after dry needling, compared to sham needling, will be assessed by the Neck Disability Index. The Neck Disability Index consists of 10 questions, each with 6 answer options with concomitant scores ranging from 0 to 5, which makes the total score of the NDI on 50. A score between 5 and 14 represents a mild disability, whereas a score between 15 and 24 is interpreted as a moderate disability. NDI scores of 25 or higher reflect a severe disability. Subjects will have to report their actual disability complaints at baseline, immediately after dry or sham needling + manual therapy and 1 week after the intervention.
Changes in headache related disability | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Changes in headache disability scores after dry needling, compared to sham needling, will be assessed by the Headache Disability Index. The Headache Disability Index consists of 25 questions which can be answered with yes (4 points), sometimes (2 points) and no (0 points). A total score of 10-28 is considered to indicate mild disability; 30-48 is moderate disability; 50-68 is severe disability; 72 or more is complete disability. Subjects will have to report their actual disability complaints at baseline, immediately after dry or sham needling + manual therapy and 1 week after the intervention.
Changes in Global Perceived Effect | immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Changes in Global Perceived Effect scores after dry needling, compared to sham needling, as assessed by the Global Perceived Effect Scale. This scale consists of 7 scores (ranging from 1 (very much better) to 7 (very much worser).
  Subjects will have to report their global perceived effect at baseline, immediately after dry or sham needling + manual therapy and 1 week after the intervention.
Changes in headache impact. | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Changes in headache impact after dry needling, compared to sham needling, as assessed by the Headache Impact Test (HIT-6) Subjects will have to report their headache impact at baseline, immediately after dry or sham needling + manual therapy and 1 week after the intervention.
Changes in global cervical mobility after dry needling or sham needling. | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Changes in global cervical mobility after dry needling or sham needling will be assessed at baseline, immediately after the intervention (needling + manual therapy) and 1 week after treatment. Measurements will be registered with the digital EasyAngle Goniometer (Meloq).
  The change in global cervical mobility will be expressed in degrees.
Change in Pain Pressure Thresholds (PPTs) | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Changes in PPTs after dry needling or sham needling will be assessed at baseline, immediately after the intervention (needling + manual therapy) and 1 week after treatment. Measurements will be registered with the digital hand-held pressure algometer (Wagner FPX 25 Force Gage). The change in PPTs will be expressed in Newton.
  To standardize the pressure applied by the investigator, the same investigator always stabilized his wrist with his other hand. The PPT assessment was performed two times with a 30-second break between each application and the pressure was increased by 1N/s until the patient reported the pressure as unpleasant. This pressure was taken as PPT expressed in Newton (N); and the average will be taken of the three measurements on the spinous process of C2 and the Upper Trapezius Muscle.
Changes in joint position error | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Changes in joint position error after dry needling or sham needling will be assessed at baseline, immediately after the intervention (needling + manual therapy) and 1 week after treatment. Measurements will be registered with the digital Motion Guidance Laser.
  The Cervical Joint Position Error (JPE) Test is a measurement tool used to clinically assess an individual's cervicocephalic proprioception ability. Cervicocephalic proprioception describes one's sense of position of their head and neck in space. The Cervical JPE Test measures the ability of a blindfolded patient to accurately relocate their head position back to a predetermined neutral point after cervical joint movement.
Motor control of the cervical spine (craniocervical flexion test) | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  The Craniocervical flexion test (CCFT) is a clinical test of neuromotor control including the activation and endurance of the deep flexors of the cervical spine. This test involves the subject performing a "yes" like nod which is the anatomical action of the Deep Cervical flexors, against a pressure biofeedback.
  Two subscores will be used: for performance and for endurance of the deep cervical flexors.
Psychosocial headache related parameters: central sensitization, pain catastrophizing, pain coping and pain related fear. | Baseline, immediately after the intervention (needling + manual therapy), 1 week after the needling intervention.
  Psychosocial related parameters: Central Sensitization Index (CSI) + Pain Catastrophizing Scale (PCS) + Pain Coping Strategies (PCI) + Pain Related Fear: Tampa Scale of Kinesiophobia (TSK)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, Prof., Principal Investigator — University Ghent
Locations (1):
- University Ghent - campus UZ Ghent - Rehabilitation Sciences B3, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No